CLINICAL TRIAL: NCT02223468
Title: Prospective Study To Characterize The Human Microbiota In Liver Transplantation And Its Impact On Early Outcome
Brief Title: Human Microbiota and Liver Transplant
Status: Completed | Type: Observational
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Cristina Dopazo Taboada, Consultant in HPB Surgery and Transplants, Hospital Vall d'Hebron
Other Study IDs: Microta.LT.14
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Intestinal Microbiota; Complication of Transplanted Liver; Acute Rejection of Liver Transplant; Infection
Keywords: Intestinal Microbiota; Liver Transplant; Acute Rejection; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples Portal nodes Periphereal blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CASE-CONTROL: CASE: Liver transplant recipients (n=20) CONTROL: A healthy person with a similar age (±10 years) to the control selected from the same family setting (n=20)

SUMMARY:
The microbiota represents the collections of microbial communities that colonize a host. In health, the microbiota protects against pathogens and maturation of the immune system. In return, the immune system determines the composition of the microbiota. Altered microbial composition (dysbiosis) has been correlated with a number of diseases in humans. The real role of the microbiota in transplant recipients is still unknown even though we suspect that it may be affected directly or indirectly by immunosuppressive drugs and antimicrobial prophylaxis taken by transplant patients, as well as by inflammatory process secondary to ischemia/reperfusion injury.

A number of studies have investigated the impact of liver transplantation on the intestinal microbiota. In a recent analysis of stool flora (Microb Ecol 2013; 65: 781-791) in 12 liver transplant recipients, changes in the microbiota were correlated to post-transplant infections. The authors suggested that the shift to pathogenic strains of bacteria due to the use of prophylactic antibiotics may be contributing to post-transplant complications. In a larger study, Wu et al (Hepatobiliary Pancreat Dis Int 2012; 11: 40-50) demonstrated marked changes in the gut microbiota post-transplantation with an increase in Enterobacteriaceae and Enterococcus, and reduction in Eubacteria, Bifidobacterium and Lactobacillus species. These changes, however, resolved over time such that by 6 months, at times when bacterial prophylaxis ends and immunosuppression is reduced.

A better characterization of the impact of post-transplant therapy on the human microbiota has the potential to improve our understanding of the infection process and translate into development of new therapeutic strategies.

The main goal of this study is to characterize intestinal microbiota and confirm the same bacterial DNA in peripheral blood and portal lymph nodes in patients affected with end-stage chronic liver disease, and to analyze its evolution from the moment of inclusion in waiting list throughout the first year after liver transplantation. For each patient, a healthy CONTROL with a similar age (± 10 years) will be selected from the same family setting, in whom just one sample will be obtained during the enrollment phase.

The second goal is to analyze the potential associations between microbiota flora and transplant outcomes during the same period.

ELIGIBILITY:
Inclusion Criteria:

* First liver transplant
* Patients aged 18-70 years
* Able to consent and agree in participate in the current study for one year

Exclusion Criteria:

* Multiorgan transplantation and/or liver transplant from cardiac arrest donor and/or with ABO incompatibility.
* Uncontrolled concomitant infections (including HIV seropositivity) and/or diarrhoea, vomiting or active gastric ulcer.
* Fulminant hepatic insufficiency as first indication for liver transplant
* Hemodynamic instability prior to liver transplant.
* Recipient presenting present or previous neoplasia, except for non-metastatic basal of squamous cutaneous carcinoma or localized hepatocarcinoma with diameter <5cm or <3known lesions with diameter <3cm.
* Significant comorbidity
* Breastfeeding or female patients at fertile age without negative pregnancy test and accepting the use of reliable fertility control method
* Any pretransplant antibiotherapy (oral or endovenous) or enrolled in any clinical assay

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult liver transplant patients in Hospital Vall d´Hebron (Barcelona, Spain)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Analyses of changes in microbiota composition before and post-transplant | Before transplant, 1st, 3rd, 7th, 14th and 28th post-transplant and 3rd, 6th, 9th and 12th months post-transplant
  Stool samples will be obtained from the liver transplant recipient following the time frame described above.
  A healthy CONTROL with a similar age (± 10 years) will be selected from the same family setting, in whom just one sample will be obtained during the enrollment phase

SECONDARY OUTCOMES:
Incidence of biopsy proven acute cellular rejection | Evaluation at 3rd, 6th, 9th and 12th months post-trasplant
  If liver dysfunction is observed, percutaneous liver biopsy will be performed and histological severity will be searching following the Banff criteria
Incidence of post-transplant infection requiring antibiotherapy (oral or endovenous) | Evaluation at 3rd, 6th, 9th and 12th months post-trasplant
Incidence of Diabetes Mellitus de novo post-transplant | 12 months post-trasplant
Incidence of Obesity (BMI≥30 kg/m2) post-transplant | 12 months post-transplant
Incidence of renal dysfunction (creatinine ≥ 1.5mg/dL and/or MDRD formula Glomerular Filtrate Rate < 60 mL/min/1.73m2) | Evaluation at 3rd, 6th, 9th and 12th months post-trasplant
Patient and graft survival rates | Evaluation at 3rd, 6th, 9th and 12th months post-trasplant

CONTACTS AND LOCATIONS:
Overall Officials: Itxarone Bilbao, PhD/MD, Principal Investigator — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); Chaysavanh Manichanh, PhD/MD, Study Chair — Physiology and Pathophysiology of the Digestive Tract, Institut de Recerca Vall d´Hebron, Barcelona (Spain); Cristina Dopazo, PhD/MD, Study Chair — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); Francisco Guarner, PhD/MD, Study Chair — Department of Gastroenterology Disease, Hospital Vall d´Hebron (Barcelona, Spain); Mireia Caralt, PhD/MD, Study Chair — Department of HBP Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); Lluis Castells, PhD/MD, Study Chair — Department of Internal Medicine, Liver Unit, Hospital Vall d´Hebron (Barcelona, Spain); Jose Luis Lazaro, MD, Study Chair — Department of HBP Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); Fernando Azpiroz, PhD/MD, Study Chair — Department of Gastroenterology Disease, Hospital Vall d´Hebron (Barcelona, Spain); Ramón Charco, PhD/MD, Study Chair — Department of HBP Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain)
Locations (1):
- Institut de Recerca Hospital Vall d´Hebron, Barcelona, Spain

REFERENCES:
- [Background] Ley RE, Peterson DA, Gordon JI. Ecological and evolutionary forces shaping microbial diversity in the human intestine. Cell. 2006 Feb 24;124(4):837-48. doi: 10.1016/j.cell.2006.02.017. PMID 16497592
- [Background] Arumugam M, Raes J, Pelletier E, Le Paslier D, Yamada T, Mende DR, Fernandes GR, Tap J, Bruls T, Batto JM, Bertalan M, Borruel N, Casellas F, Fernandez L, Gautier L, Hansen T, Hattori M, Hayashi T, Kleerebezem M, Kurokawa K, Leclerc M, Levenez F, Manichanh C, Nielsen HB, Nielsen T, Pons N, Poulain J, Qin J, Sicheritz-Ponten T, Tims S, Torrents D, Ugarte E, Zoetendal EG, Wang J, Guarner F, Pedersen O, de Vos WM, Brunak S, Dore J; MetaHIT Consortium; Antolin M, Artiguenave F, Blottiere HM, Almeida M, Brechot C, Cara C, Chervaux C, Cultrone A, Delorme C, Denariaz G, Dervyn R, Foerstner KU, Friss C, van de Guchte M, Guedon E, Haimet F, Huber W, van Hylckama-Vlieg J, Jamet A, Juste C, Kaci G, Knol J, Lakhdari O, Layec S, Le Roux K, Maguin E, Merieux A, Melo Minardi R, M'rini C, Muller J, Oozeer R, Parkhill J, Renault P, Rescigno M, Sanchez N, Sunagawa S, Torrejon A, Turner K, Vandemeulebrouck G, Varela E, Winogradsky Y, Zeller G, Weissenbach J, Ehrlich SD, Bork P. Enterotypes of the human gut microbiome. Nature. 2011 May 12;473(7346):174-80. doi: 10.1038/nature09944. Epub 2011 Apr 20. PMID 21508958
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Wells JM, Rossi O, Meijerink M, van Baarlen P. Epithelial crosstalk at the microbiota-mucosal interface. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4607-14. doi: 10.1073/pnas.1000092107. Epub 2010 Sep 8. PMID 20826446
- [Background] Seki E, Schnabl B. Role of innate immunity and the microbiota in liver fibrosis: crosstalk between the liver and gut. J Physiol. 2012 Feb 1;590(3):447-58. doi: 10.1113/jphysiol.2011.219691. Epub 2011 Nov 28. PMID 22124143
- [Background] Guarner F, Malagelada JR. Gut flora in health and disease. Lancet. 2003 Feb 8;361(9356):512-9. doi: 10.1016/S0140-6736(03)12489-0. PMID 12583961
- [Background] O'Hara AM, Shanahan F. Gut microbiota: mining for therapeutic potential. Clin Gastroenterol Hepatol. 2007 Mar;5(3):274-84. doi: 10.1016/j.cgh.2006.12.009. PMID 17368226
- [Background] Neufeld KM, Kang N, Bienenstock J, Foster JA. Reduced anxiety-like behavior and central neurochemical change in germ-free mice. Neurogastroenterol Motil. 2011 Mar;23(3):255-64, e119. doi: 10.1111/j.1365-2982.2010.01620.x. Epub 2010 Nov 5. PMID 21054680
- [Background] Maynard CL, Elson CO, Hatton RD, Weaver CT. Reciprocal interactions of the intestinal microbiota and immune system. Nature. 2012 Sep 13;489(7415):231-41. doi: 10.1038/nature11551. PMID 22972296
- [Background] Guarner F, Bourdet-Sicard R, Brandtzaeg P, Gill HS, McGuirk P, van Eden W, Versalovic J, Weinstock JV, Rook GA. Mechanisms of disease: the hygiene hypothesis revisited. Nat Clin Pract Gastroenterol Hepatol. 2006 May;3(5):275-84. doi: 10.1038/ncpgasthep0471. PMID 16673007
- [Background] Oh PL, Martinez I, Sun Y, Walter J, Peterson DA, Mercer DF. Characterization of the ileal microbiota in rejecting and nonrejecting recipients of small bowel transplants. Am J Transplant. 2012 Mar;12(3):753-62. doi: 10.1111/j.1600-6143.2011.03860.x. Epub 2011 Dec 7. PMID 22152019
- [Background] Xie Y, Luo Z, Li Z, Deng M, Liu H, Zhu B, Ruan B, Li L. Structural shifts of fecal microbial communities in rats with acute rejection after liver transplantation. Microb Ecol. 2012 Aug;64(2):546-54. doi: 10.1007/s00248-012-0030-1. Epub 2012 Mar 21. PMID 22430504
- [Background] Wu ZW, Ling ZX, Lu HF, Zuo J, Sheng JF, Zheng SS, Li LJ. Changes of gut bacteria and immune parameters in liver transplant recipients. Hepatobiliary Pancreat Dis Int. 2012 Feb;11(1):40-50. doi: 10.1016/s1499-3872(11)60124-0. PMID 22251469
- [Background] Rayes N, Seehofer D, Theruvath T, Schiller RA, Langrehr JM, Jonas S, Bengmark S, Neuhaus P. Supply of pre- and probiotics reduces bacterial infection rates after liver transplantation--a randomized, double-blind trial. Am J Transplant. 2005 Jan;5(1):125-30. doi: 10.1111/j.1600-6143.2004.00649.x. PMID 15636620
- [Background] Fricke WF, Maddox C, Song Y, Bromberg JS. Human microbiota characterization in the course of renal transplantation. Am J Transplant. 2014 Feb;14(2):416-27. doi: 10.1111/ajt.12588. Epub 2013 Dec 26. PMID 24373208
- [Background] Alegre ML, Mannon RB, Mannon PJ. The microbiota, the immune system and the allograft. Am J Transplant. 2014 Jun;14(6):1236-48. doi: 10.1111/ajt.12760. Epub 2014 May 19. PMID 24840316
- [Background] Lu H, He J, Wu Z, Xu W, Zhang H, Ye P, Yang J, Zhen S, Li L. Assessment of microbiome variation during the perioperative period in liver transplant patients: a retrospective analysis. Microb Ecol. 2013 Apr;65(3):781-91. doi: 10.1007/s00248-013-0211-6. Epub 2013 Mar 17. PMID 23504024